CLINICAL TRIAL: NCT04563416
Title: Application of Artificial Intelligence for Early Diagnosis of Gastric Cancer During Optical Enhancement Magnifying Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2018SDU-QILU-3
Record Dates: First submitted 2020-09-22; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Artificial Intelligence; Optical Enhancement Endoscopy; Magnifying Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who need undergo magnifying endoscopy

SUMMARY:
Previous prospective randomized controlled study demonstrated higher accuracy rate of diagnosing early gastric cancers by Magnifying image-enhanced endoscopy than conventional white-light endoscopy. Nevertheless, it is difficult to differentiate early gastric cancer from noncancerous lesions for beginner. we developed a new computer-aided system to assist endoscopists in identifying early gastric cancers in magnifying optical enhancement images.

DETAILED DESCRIPTION:
Gastric cancer is the third most common cause of cancer-associated deaths worldwide especially in Asia.Early detection and treatment would cure the disease with 5-year survival rate greater than 90%.However, the sensitivity of conventional endoscopy with white-light imaging (C-WLI) in diagnosis of early gastric cancers (EGCs) is merely 40%. Magnifying image-enhanced endoscopy (IEE) techniques such as magnifying narrow band imaging (M-NBI) have been developed and 2 RCT report that white-light imaging combine with M-NBI can increase the sensitivity to 95%. The strategy that using white-light imaging to detect the suspicious lesion and using M-IEE techniques to make a diagnosis of early gastric cancer is recommend in screening endoscopy.

Optical enhancement (OE) which is one of the M-IEE techniques was developed by HOYA Co. (Tokyo, Japan) . This technology combines digital signal processing and optical filterers to clear display of mucosal microsurface (MS) and microvessel (MV). The advantage of OE is to overcome the darkness of NBI which leads to less usefulness for detect-ability in the full extended gastrointestinal lumen.Nevertheless, it is difficult to differentiate early gastric cancer from noncancerous lesions for beginner, and expertise with sub-optimal inter-observer agreement is essential for the use of M-IEE.

Nowadays, Artificial intelligence (AI) using deep machine learning has made a major breakthrough in gastroenterology, which using gradient descent method and backpropagation to automatically extract specific images features. The diagnostic accuracy in identifying upper gastrointestinal cancer was 0.955 in C-WLI . Polyps can be identified in real time with 96% accuracy in screening colonoscopy. AI show an outstanding application in detection and diagnosis.

This study aims to develop a M-OE assistance model in the diagnosis of EGCs by distinguishing cancer or not.

ELIGIBILITY:
Inclusion Criteria:

* patients receive optical magnifying OE endoscopy examination

Exclusion Criteria:

* Patients with advanced cancer, lymphoma,active stage of ulcer and artificial ulcer after ESD were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients suspected of early gastric cancer and receive optical magnifying OE endoscopy examination.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
the diagnosis efficiency of the computer-assist diagnosis tool | 12 months
  the sensitivity, specificity and accuracy of the computer-assist diagnosis tool

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PHD, Principal Investigator — Study Principal Investigator Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Ma M, Li Z, Yu T, Liu G, Ji R, Li G, Guo Z, Wang L, Qi Q, Yang X, Qu J, Wang X, Zuo X, Ren H, Li Y. Application of deep learning in the real-time diagnosis of gastric lesion based on magnifying optical enhancement videos. Front Oncol. 2022 Aug 5;12:945904. doi: 10.3389/fonc.2022.945904. eCollection 2022. PMID 35992850